CLINICAL TRIAL: NCT01627782
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Group, Dose Frequency Study of Ketamine in Subjects With Treatment-resistant Depression
Brief Title: A Study of Ketamine in Patients With Treatment-resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR100886; KETIVTRD2002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Treatment-resistant depression; Ketamine
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (4):
- Placebo 3 times/week (Placebo Comparator)
  Interventions: Drug: Placebo
- Ketamine 3 times/week (Experimental)
  Interventions: Drug: Ketamine
- Ketamine 2 times/week (Experimental)
  Interventions: Drug: Ketamine
- Placebo 2 times/week (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Form= intravenous infusion, route= intravenous (IV) use. IV infusions of placebo 2 times weekly or IV infusions of placebo 3 times weekly.
  Arms: Placebo 2 times/week; Placebo 3 times/week
Drug: Ketamine — Type= exact number, unit= mg/kg, number= 0.5, form= intravenous infusion, route= intravenous (IV) use. IV infusions of ketamine 0.50 mg/kg, 2 times weekly or IV infusions of ketamine 0.50 mg/kg, 3 times weekly.
  Arms: Ketamine 2 times/week; Ketamine 3 times/week

SUMMARY:
The purpose of this study is to explore the optimal dose frequency of ketamine in patients with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This is a double-blind (patients and study personnel do not know the identity of the administered treatments), randomized (the drug is assigned by chance), placebo-controlled (placebo is a substance that appears identical to the treatment and has no active ingredients), parallel arm study (each group of patients will be treated at the same time). The study will consist of a screening phase of up to 4 weeks, a 4-week double-blind treatment phase (Day 1 to Day 29), and a 3-week post treatment (follow up) phase. In the double-blind phase, patients will receive over 4 weeks either intravenous (IV) infusions of placebo (2 or 3 times weekly) or IV infusions of ketamine (2 or 3 times weekly). The total study duration for each patient will be a maximum of 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Be medically stable on the basis of clinical laboratory tests performed at screening
* Meet diagnostic criteria for recurrent major depressive disorder (MDD), without psychotic features
* Have a history of inadequate response, ie treatment was not successful, to at least 1 antidepressant
* Have an Inventory of Depressive Symptoms-Clinician rated, 30 item (IDS-C30) total score >= 40 at screening and predose at Day 1
* Inpatient or agreed to be admitted to the clinic on each dosing day

Exclusion Criteria:

* Has uncontrolled hypertension
* Has a history of, or current signs and symptoms of diseases, infections or conditions that in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the patient or that could prevent, limit, or confound the protocol-specified assessments
* Has known allergies, hypersensitivity, or intolerance to ketamine or its excipients
* Is unable to read and understand the consent forms and patient reported outcomes, complete study-related procedures, and/or communicate with the study staff

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2012-08-06 (Actual); Primary Completion 2013-09-12 (Actual); Study Completion 2013-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (13):
- United States (13):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Centennial, Colorado
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Atlanta, Georgia
  - Rockville, Maryland
  - Marlton, New Jersey
  - New York, New York
  - Allentown, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah

REFERENCES:
- [Derived] Lewis S, Romano C, De Bruecker G, Murrough JW, Shelton R, Singh JB, Jamieson C. Analysis of Clinical Trial Exit Interview Data in Patients with Treatment-Resistant Depression. Patient. 2019 Oct;12(5):527-537. doi: 10.1007/s40271-019-00369-8. PMID 31270774
- [Derived] Johnson KM, Devine JM, Ho KF, Howard KA, Saretsky TL, Jamieson CA. Evidence to Support Montgomery-Asberg Depression Rating Scale Administration Every 24 Hours to Assess Rapid Onset of Treatment Response. J Clin Psychiatry. 2016 Dec;77(12):1681-1686. doi: 10.4088/JCP.15m10253. PMID 28086004
- See also: A Double-blind, Randomized, Placebo-controlled, Parallel Group, Dose Frequency Study of Ketamine in Subjects With Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR100886&attachmentIdentifier=7d6ebba0-1b0a-4df6-96fd-421b53fdb5b7&fileName=KETIVTRD2002_(CR100886)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 165 participants were screened and 68 participants were randomized into the study. Of these 68 participants randomized, 67 participants received at least 1 dose of the study agent (Intent-To-Treat analysis set).
Groups:
- Placebo: 2 Times Per Week: Participants received Intravenous (IV) infusion of placebo 2 times weekly for 4 weeks.
- Ketamine: 2 Times Per Week: Participants received 0.50 milligram per kilogram (mg/kg) ketamine IV infusion 2 times weekly for 4 weeks.
- Placebo: 3 Times Per Week: Participants received IV infusion of placebo 3 times weekly for 4 weeks.
- Ketamine: 3 Times Per Week: Participants received 0.50 mg/kg ketamine IV infusion 3 times weekly for 4 weeks.
Period: Overall Study
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Started | 17 | 18 | 16 | 17
Treated | 16 | 18 | 16 | 17
Completed | 1 | 12 | 1 | 11
Not Completed | 16 | 6 | 15 | 6
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 11 | 1 | 15 | 2
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 3
Not completed — Randomized But Not Treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat (ITT) analysis set is defined as participants who were randomized and received at least 1 dose of the study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week | Total
Number analyzed (Participants) | 16 | 18 | 16 | 17 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.79) | 45.7 (9.58) | 46.1 (10.51) | 43.3 (11.99) | 43.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 9 | 12 | 45
  Male | 4 | 6 | 7 | 5 | 22
Region of Enrollment [Number; unit: participants]
  USA | 16 | 18 | 16 | 17 | 67

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Day 15
Description: The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Time Frame: Baseline (Day 1) and Day 15
Population: An intent-to-treat (ITT) analysis set is defined as all participants who receive at least 1 dose of study drug and have both Day 1 (baseline) and at least 1 post-baseline MADRS total score. Here,"N"(Number of Participants Analyzed) and "n" signifies those participants who were evaluable for this outcome measure and at given time point, respectively
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 18 | 16 | 17
Units on a scale
  Baseline (n=16,18,16,17) | 35.6 (3.79) | 33.3 (4.91) | 36.8 (5.83) | 35.4 (5.28)
  Change at Day 15 (n=13,16,16,13) | -5.7 (10.23) | -18.4 (12.01) | -3.1 (5.67) | -17.7 (7.27)
Statistical Analysis 1: Comparison: Placebo: 2 Times Per Week vs Ketamine: 2 Times Per Week; Test type: Superiority or Other; p < 0.001, Mixed Effect Model Repeated Measure; Difference of Least Square Means = -16.0, 70% CI 2-sided [-20.00 to -12.01]
Statistical Analysis 2: Comparison: Placebo: 3 Times Per Week vs Ketamine: 3 Times Per Week; Test type: Superiority or Other; p < 0.001, Mixed Effect Model Repeated Measure; Difference of Least Square Means = -16.4, 70% CI 2-sided [-18.96 to -13.84]

2. Secondary Outcome: Change in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score From Baseline to Day 29
Description: as for outcome 1
Time Frame: Baseline (Day 1) and Day 29
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 18 | 16 | 17
Units on a scale
  Baseline (n=16,18,16,17) | 35.6 (3.79) | 33.3 (4.91) | 36.8 (5.83) | 35.4 (5.28)
  Change at Day 29 (n=2,13,1,13) | -23.5 (10.61) | -27.1 (6.60) | -1 (NA) — Standard deviation was not evaluable since only 1 participant was evaluated. | -22.9 (10.61)

3. Secondary Outcome: Number of Responders Based on Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Participants with a reduction in the MADRS total score of greater than or equal to (>=) 50 percent from baseline were defined as responders. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Time Frame: Day 15 and Day 29
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 16 | 16 | 13
Participants
  Day 15 (n=13,16,16,13) | 2 (3.79) | 11 (4.91) | 1 (5.83) | 7 (5.28)
  Day 29 (n=2,13,1,13) | 1 (10.61) | 13 (6.60) | 0 (NA) | 9 (10.61)

4. Secondary Outcome: Number of Remitters Based on Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Participants who had a MADRS total score of less than or equal to (<=) 10 were considered remitters. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Time Frame: Day 15 and Day 29
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 16 | 16 | 13
Participants
  Day 15 (n=13,16,16,13) | 1 (3.79) | 6 (4.91) | 0 (5.83) | 3 (5.28)
  Day 29 (n=2,13,1,13) | 1 (10.61) | 12 (6.60) | 0 (NA) | 5 (10.61)

5. Secondary Outcome: Number of Sustained Responders Based on Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Sustained response on Day 15 was defined as achieving an onset of antidepressant response within the first week that is maintained to the end of study Day 15. The MADRS is a clinician-rated scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher scores represent a more severe condition.
Time Frame: Day 15
Population: An intent-to-treat (ITT) analysis set is defined as all participants who receive at least 1 dose of study drug and have both Day 1 (baseline) and at least 1 post-baseline MADRS total score. Here, "N" (Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 18 | 16 | 17
Participants | 1 (3.79) | 7 (4.91) | 0 (5.83) | 4 (5.28)

6. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Score From Baseline to Endpoint (Day 29)
Description: The CGI-S was used to rate the severity of the participants illness at the time of assessment, relative to the clinician's past experience with participants who had the same diagnosis and improvement with treatment. Considering total clinical experience, a participant was assessed on severity of mental illness at the time of rating according to: 0= not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants.
Time Frame: Baseline (Day 1) and Endpoint (Day 29)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 15 | 18 | 16 | 17
Units on a scale
  Baseline (n=15,18,16,17) | 5.0 (3.79) [4 to 6] | 5.0 (4.91) [4 to 6] | 5.0 (5.83) [4 to 6] | 5.0 (5.28) [4 to 6]
  Change at Endpoint (n=15,18,16,17) | 0.0 (10.61) [-4 to 0] | -2.0 (6.60) [-4 to 1] | 0.0 (NA) [-1 to 1] | -2.0 (10.61) [-4 to 0]

7. Secondary Outcome: Clinical Global Impression of Improvement (CGI-I) Score at Endpoint of Double Blind Phase
Description: The CGI-I is a 7-point scale that was used to assess how much the participants illness was improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 0= not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse.
Time Frame: Endpoint (Day 29)
Population: An intent-to-treat (ITT) analysis set is defined as all participants who receive at least 1 dose of study drug and have both Day 1 (baseline) and at least 1 post-baseline MADRS total score. Here,"N"(Number of Participants Analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 18 | 16 | 17
Units on a scale | 4.0 (3.79) [1 to 5] | 2.0 (4.91) [1 to 5] | 4.0 (5.83) [2 to 5] | 2.0 (5.28) [1 to 5]

8. Secondary Outcome: Change in Patient Global Impression-Severity (PGI-S) Score From Baseline to Endpoint (Day 29)
Description: The PGI-S is an 11-point (0 to 10) scale that required the participant to rate the severity of their illness at the time of assessment, relative to the participants past experience. Considering their total experience, the participant was to assess the severity of their depression illness at the time of rating as none, mild, moderate or severe. The scale is rated as, 0=very well and 10=very poor.
Time Frame: Baseline (Day 1) and Endpoint (Day 29)
Population: as for outcome 1
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 15 | 18 | 16 | 17
Units on a scale
  Baseline (n=15,18,16,17) | 8.0 (3.79) [4 to 9] | 7.5 (4.91) [5 to 9] | 8.0 (5.83) [5 to 10] | 7.0 (5.28) [5 to 9]
  Change at Endpoint (n=15,18,16,17) | 0.0 (10.61) [-3 to 2] | -4.0 (6.60) [-8 to 0] | -1.0 (NA) [-3 to 1] | -3.0 (10.61) [-8 to 1]

9. Secondary Outcome: Patient Global Impression-Change (PGI-C) Score at Endpoint of Double Blind Phase
Description: The PGI-C is a 7-point scale that required the subject to assess how much their illness had improved or worsened relative to a baseline state at the beginning of the intervention. The response options were: very much improved; much improved; improved (just enough to make a difference); no change; worse (just enough to make a difference); much worse; or very much worse. The scale is rated as, 1=very much improved and 7=very much worse.
Time Frame: Endpoint (Day 29)
Population: as for outcome 7
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 18 | 16 | 17
Units on a scale | 4.0 (3.79) [2 to 6] | 2.0 (4.91) [1 to 4] | 4.0 (5.83) [3 to 6] | 3.0 (5.28) [1 to 4]

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ketamine
Description: The Cmax is the maximum observed plasma concentration of drug.
Time Frame: Pre-infusion, 20, 40 (End of the Infusion), 45, 50, 60, 90, 120, 180, 240 and 360 minutes post-infusion on Day 1 and Day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/ml)
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 16
nanogram per milliliter (ng/ml)
  Day 1 (n=16,16) | 207 (83.0) [5 to 9] | 168 (34.4) [5 to 9]
  Day 15 (n=14,15) | 219 (69.4) [-8 to 0] | 189 (74.4) [-8 to 1]

11. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Ketamine
Description: The Tmax is defined as actual sampling time to reach maximum observed drug concentration.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Median (Full Range); unit: Hour
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 16
Hour
  Day 1 (n=16,16) | 0.67 (83.0) [0.63 to 0.83] | 0.66 (34.4) [0.33 to 0.75]
  Day 15 (n=14,15) | 0.67 (69.4) [0.63 to 1.00] | 0.67 (74.4) [0.5 to 0.83]

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC[0-last])
Description: The AUC(0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 16 | 15
hour*nanogram per milliliter
  Day 1 (n=16,15) | 312 (67.9) [0.63 to 0.83] | 295 (42.8) [0.33 to 0.75]
  Day 15 (n=14,14) | 342 (66.7) [0.63 to 1.00] | 293 (65.6) [0.5 to 0.83]

13. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity])
Description: The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 13
hour*nanogram per milliliter
  Day 1 (n=13,13) | 369 (79.9) [0.63 to 0.83] | 344 (47.3) [0.33 to 0.75]
  Day 15 (n=9,8) | 416 (68.9) [0.63 to 1.00] | 340 (94.0) [0.5 to 0.83]

14. Secondary Outcome: Total Systemic Clearance (CL) of Ketamine
Description: The CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 13
liter per hour
  Day 1 (n=13,13) | 113 (35.1) [0.63 to 0.83] | 108 (21.4) [0.33 to 0.75]
  Day 15 (n=9,8) | 93.9 (15.6) [0.63 to 1.00] | 117 (22.3) [0.5 to 0.83]

15. Secondary Outcome: Volume of Distribution at Steady-State (Vss) of Ketamine
Description: The Vss is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of ketamine at steady state.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 13
liter
  Day 1 (n=13,13) | 275 (114) [0.63 to 0.83] | 276 (77.2) [0.33 to 0.75]
  Day 15 (n=9,8) | 239 (61.2) [0.63 to 1.00] | 290 (64.9) [0.5 to 0.83]

16. Secondary Outcome: Elimination Half-Life (t1/2)
Description: The elimination half-life (t1/2) is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Ketamine: 2 Times Per Week | Ketamine: 3 Times Per Week
Number analyzed (Participants) | 13 | 13
hour
  Day 1 (n=13,13) | 2.18 (0.43) [0.63 to 0.83] | 2.18 (0.40) [0.33 to 0.75]
  Day 15 (n=9,8) | 2.39 (0.36) [0.63 to 1.00] | 2.21 (0.36) [0.5 to 0.83]

ADVERSE EVENTS:
Time Frame: Screening up to Follow up (3 Weeks After Last Dose of Study Drug Administration)
Description: The safety analysis set is defined as all participants who received at least 1 dose of the study drug.
Arm/Group | Placebo: 2 Times Per Week | Ketamine: 2 Times Per Week | Placebo: 3 Times Per Week | Ketamine: 3 Times Per Week
Serious Adverse Events (participants affected / at risk) | 0/16 | 2/18 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 9/16 | 15/18 | 8/16 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: 2 Times Per Week (N=16) | Ketamine: 2 Times Per Week (N=18) | Placebo: 3 Times Per Week (N=16) | Ketamine: 3 Times Per Week (N=17)
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo: 2 Times Per Week (N=16) | Ketamine: 2 Times Per Week (N=18) | Placebo: 3 Times Per Week (N=16) | Ketamine: 3 Times Per Week (N=17)
Cardiac Flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Altered Visual Depth Perception (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 1 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 2 | 4
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 2
Feeling Abnormal (General disorders) | 0 | 1 | 0 | 1
Feeling Cold (General disorders) | 0 | 0 | 0 | 1
Inflammation (General disorders) | 0 | 1 | 0 | 0
Infusion Site Pain (General disorders) | 0 | 1 | 0 | 1
Injection Site Extravasation (General disorders) | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0 | 0
Groin Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Blood Potassium Decreased (Investigations) | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 2 | 0 | 0
Drug Screen Positive (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram St-T Change (Investigations) | 0 | 0 | 0 | 1
Weight Decreased (Investigations) | 0 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 4 | 0 | 2
Dizziness Postural (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 5 | 4 | 1 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 0 | 3
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 2
Poor Quality Sleep (Nervous system disorders) | 0 | 1 | 0 | 0
Sedation (Nervous system disorders) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 4 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Dissociation (Psychiatric disorders) | 0 | 5 | 0 | 1
Dissociative Disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Euphoric Mood (Psychiatric disorders) | 0 | 1 | 0 | 1
Hallucination, Tactile (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination, Visual (Psychiatric disorders) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition Urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.